CLINICAL TRIAL: NCT03823781
Title: Prophylactic Milrinone Infusion for the Prevention Low Cardiac Output Syndrome After Corrective Surgery for Congenital Heart Disease in Infants: A Randomized, Multi-center, Double-blinded, Placebo-controlled Study
Brief Title: Prophylactic Use of Milrinone After Congenital Heart Surgery in Infants
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCMCIRB-K2018105
Record Dates: First submitted 2019-01-25; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Low Cardiac Output Syndrome; Cardiac Surgical Procedures; Infant
MeSH Terms: conditions — Cardiac Output, Low | interventions — Milrinone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- milrinone (Experimental): milrinone milrinone will be administered intravenously at a rate of 0.75ug/kg/min for 35 hours, and baseline catecholamines will be administered at the discretion of the physician.
  Interventions: Drug: Milrinone
- normal saline (Placebo Comparator): placebo placebo (normal saline) will be administered intravenously for 35 hours, and baseline catecholamines will be administered at the discretion of the physician.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Milrinone — The study intervention is an intravenous infusion of milrinone or placebo.
  Other Names: Milrinone Lactate
  Arms: milrinone
Drug: Normal saline — The study intervention is an intravenous infusion of milrinone or placebo.
  Other Names: Normal Saline 0.9% Infusion Solution Bag
  Arms: normal saline

SUMMARY:
This randomized, multi-center, double-blinded, placebo-controlled study is designed to evaluate the efficacy and safety of milrinone compared with placebo in participants after corrective surgery for congenital heart disease. Participants will be randomized in a 1:1 ratio within 90 minutes after arriving in the intensive care unit (ICU), to receive either intravenous milrinone or placebo for 36 hours. Participants will be stratified according Vasoactive Inotrope Score after arriving in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Age younger than 12 months
* Without pre-operative low cardiac output syndrome
* Bi-ventricular repair of congenital heart disease involving cardiopulmonary bypass
* Informed consent obtained from each participant's parent or guardian

Exclusion Criteria:

* A body weight <2 kg
* Prematurity (birth <36 weeks postconceptual age)
* Renal dysfunction ( Creatinine>1.5mg/dL 48 hours before surgery)
* Low cardiac output syndrome or hypotension on arrival to ICU from OR
* Cardiopulmonary resuscitation before surgery
* Platelet count<80,000/mm3 before surgery
* Left ventricular outflow tract obstruction before surgery
* Ventricular arrhythmia before surgery
* Without femoral artery catheter before arriving in the ICU
* Consent was withdrawn by participants' parent or guardian.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 520 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants died within 30 days postoperatively | up to 30 days postoperatively
Number of participants developed low cardiac output syndrome within the first 36 hours after initiation of study drug | 36 hours after initiation of study drug
  Low cardiac output syndrome was defined as the following: clinical signs or symptoms (eg, tachycardia, oliguria, poor perfusion, or cardiac arrest) with or without a widened arterial-mixed venous oxygen saturation difference or metabolic acidosis; mechanical support of the circulation (eg, extracorporeal life support, ventricular assist device), a cardiac index determined by Pulse indicator continuous cardiac output (PiCCO) of <2.2 L/min/m2

SECONDARY OUTCOMES:
Number of participants developed low cardiac output syndrome in the interval between 36 hours after initiation of study drug and the final Follow up. Cardiac index will be determined by Doppler echocardiography | up to 30 days postoperatively
Change in Vasoactive Inotrope Score. | 36 hours after initiation of study drug
  Vasoactive Inotrope Score=100*Epinephrine dose (ug/kg/min)+100*Norepinephrine dose (ug/kg/min)+10*Dopamine dose (ug/kg/min)+10*Dobutamine dose (ug/kg/min) +10,000*Vasopressin dose (units/kg/min) +10*Milrinone dose (ug/kg/min)
Length of intensive care stay. | up to 30 days postoperatively or until ICU discharge.
  Length of intensive care stay will be calculated from date of ICU admission to date of ICU discharge
Length of hospital stay. | up to 30 days postoperatively or until hospital discharge
  Length of hospital stay will be calculated from date of hospital admission to date of hospital discharge
Duration of mechanical ventilation. | up to 30 days postoperatively or until extubation
  Duration of mechanical ventilation will be calculated from date and time of ICU admission to date and time of extubation
Number of participants with improvement of ventriculoarterial coupling | 36 hours after initiation of study drug
  ventriculoarterial coupling improvement will be assessed by means of ventriculoarterial coupling values shift closer to 1. ventriculoarterial coupling will be obtained as : (1-EF)/EF
Number of participants requiring mechanical circulatory support. | up to 30 days postoperatively
  eg. Extra-Corporeal Membrane Oxygenation, ventricular assist device
Number of participants with a decrease in regional tissue oxygenation at least 20% from baseline. | 36 hours after initiation of study drug
  Cerebral and abdominal regional tissue oxygenation will be monitored
Number of participants with treatment-related adverse events | 36 hours after initiation of study drug
  Treatment-related adverse events will be evaluated by sponsor's drug safety surveillance reviewer

CONTACTS AND LOCATIONS:
Overall Officials: Huiwen Chen, MD, PhD, Study Director — Department of clinical research, Shanghai children's medical center
Locations (1):
- Shanghai Shanghai Children's Medical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided